CLINICAL TRIAL: NCT02644356
Title: Palliative Care Provider Online Education in Evidence-Based Complementary Therapies
Brief Title: Complementary Therapies in Palliative Care
Acronym: CTPC
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Collinge and Associates, Inc. (Other)
Collaborators: Kozak & Associates, LLC (Unknown)
Responsible Party: Principal Investigator, William Collinge, PhD, President, Collinge and Associates, Inc.
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: R43CA157005 (NIH)
Record Dates: First submitted 2015-12-12; First posted 2015-12-31 (Estimated); Results first posted 2017-03-17 (Actual); Last update posted 2017-03-17 (Actual); Status verified 2017-01

CONDITIONS: Health Care Provider Education

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Online CE/CME course (Experimental): Participant in taking the three course modules and completing pre- and post-course data collection.
  Interventions: Behavioral: Online CE/CME course

INTERVENTIONS:
Behavioral: Online CE/CME course — Educational modules of a proposed online CE/CME course, module topics consisting of acupuncture, massage, and music-related interventions

SUMMARY:
Palliative care represents one of the most rapidly expanding sectors of health care. Its rapid growth has been accompanied by widespread needs for training of multidisciplinary personnel to work with the unique set of health issues specific to its population of patients - not only those at end-of-life, but also patients with long-term, incurable, chronic and degenerative illnesses. This project will develop the first online continuing education program for palliative care personnel in the evidence-based application of complementary therapies, to enhance patient care and quality of life in the palliative care setting.

DETAILED DESCRIPTION:
Palliative care represents one of the most rapidly expanding sectors of health care. Its rapid growth has been accompanied by widespread needs for training of multidisciplinary personnel to work with the unique set of health issues specific to its population of patients - not only those at end-of-life, but also patients with long-term, incurable, chronic and degenerative illnesses. Selected complementary therapies offer significant benefits for reducing suffering and improving quality of life in palliative care patients; however, there currently are no systematic educational offerings on the evidence-based application of such therapies in the palliative care setting. This project will develop the first online continuing education program for palliative care personnel in the evidence-based application of complementary therapies in the palliative care setting. The final product will consist of an interactive course with eight modules; Phase I will develop the web infrastructure for the course, and will then pilot test two modules to establish feasibility of the concept. The specific aims are as follows: Aim 1. Build a website capable of delivering an online interactive educational curriculum. Aim 2. Conduct evidence-based reviews of the literature on the application of complementary therapies to pain and dyspnea in palliative care settings. Aim 3. Incorporate the course content into a structure and form that can be effectively delivered over the website. Aim 4. Conduct peer review evaluation of content to determine fidelity of course content with available evidence. Aim 5. Recruit a multidisciplinary sample of health care personnel practicing in the field of palliative care. Aim 6. Conduct pilot testing of two modules of the program. Aim 7. Evaluate {attitudinal and} learning outcomes and user satisfaction feedback to determine feasibility of the approach. Feasibility of the approach will be determined by success in recruitment, compliance, evidence of meeting user learning objectives, and user satisfaction data. The final product to be developed is an eight-module online educational course for multidisciplinary health professionals in the evidence-based application of complementary therapies in palliative care. Commercial application will be as a continuing education program that is licensed to institutions (care facilities, hospitals, universities, colleges) as well as purchased by individual users (fee-based), with discipline-specific continuing education credits available, all administered over the internet. Impact and Innovation: This will be the first online educational program for palliative care personnel on this topic available in the US. The course will spearhead the expansion of the existing paradigm of palliative care to incorporate evidence-based integration of complementary therapies. Technological innovation includes the employment of fluid updating of content to licensees, which is a new development in online education and particularly important given the rapid rate of emergence of new data. Public health benefit: The course will aid in the improvement of quality of palliative care, benefitting potentially millions of recipients in the most rapidly expanding sector of the health care system.

ELIGIBILITY:
Inclusion Criteria:

* Physicians (MD, DO), physician assistant (PA), nurse practitioner (NP), registered nurse (RN), licensed practical nurse (LPN), social worker (BA/BS/BSW, MSW, PhD/DSW), psychologist (MS/MA, PhD/PsyD), counselor (MS/MA),administrator, and chaplain.
* Must be currently active within palliative care settings.

Exclusion Criteria:

* Professionals not actively working in palliative care settings

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2011-07; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: William B Collinge, PhD, MPH, Principal Investigator — Collinge and Associates, Inc.

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Online CE/CME Course
Started | 51
Completed | 49 (49 of the 51 consented subjects completed pre-post knowledge testing (96%))
Not Completed | 2
Not completed — Withdrawal by Subject | 2

BASELINE CHARACTERISTICS:
Arm/Group | Online CE/CME Course
Number analyzed (Participants) | 51
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 51
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.8 (12.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 44
  Male | 7
Race/Ethnicity, Customized [Number; unit: participants]
  White non-hispanic | 29
  Asian American | 8
  Hispanic | 7
  Black | 6
  American Indian | 1
Region of Enrollment [Number; unit: participants]
  United States | 51

OUTCOME MEASURES:

1. Primary Outcome: Change in Test Scores on Knowledge of Course Content From Baseline to 30 Days
Description: Investigator-generated test of change in knowledge about theory, mechanisms of action, delivery, indications for use, evidence of efficacy; total of 45 multiple choice questions covering three modalities: acupuncture, massage, and music interventions. Range of total possible correct responses was from 0-45, with subscores as follows: range for acupuncture, 0-15; massage, 0-16; music interventions, 0-14. Total score is the sum of the combined subscores.
Time Frame: Baseline, 30 days
Population: Disciplines: Nursing, 22; physician, 11; social work, 13; chaplaincy, 4; administrators, 4; counseling/psychology, 2 (some reported more than one discipline).
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Online CE/CME Course
Number analyzed (Participants) | 49
units on a scale | 39.3 (6.0)

2. Secondary Outcome: Change in Ratings of Confidence in Understanding a Modality's Safety Considerations in PC From Baseline to 30 Days
Description: Investigator-generated scale of confidence in understanding modality safety considerations. Likert-scaled items ranging from 0-10, with 0 as lowest and 10 as highest.
Time Frame: Baseline, 30 days
Population: There was missing data for one subject for this item.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Online CE/CME Course
Number analyzed (Participants) | 48
units on a scale | 9.2 (1.6)

3. Secondary Outcome: Change in Ratings of Confidence in Making Evidence-based Recommendations for the Modality in PC Planning From Baseline to 30 Days
Description: Investigator-generated scale of confidence in making evidence-based recommendations about the modality. Likert-scaled items ranging from 0-10, with 0 as lowest and 10 as highest.
Time Frame: Baseline, 30 days
Population: There was missing data for one subject for this item.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Online CE/CME Course
Number analyzed (Participants) | 48
units on a scale | 9.4 (1.3)

4. Secondary Outcome: Change in Ratings of Confidence in Explaining the Modality From Baseline to 30 Days
Description: Investigator-generated scale of confidence in communicating about the modality to patients, families and colleagues in PC contexts. Likert-scaled items ranging from 0-10, with 0 as lowest and 10 as highest.
Time Frame: Baseline, 30 days
Population: There was missing data for one subject for this item.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Online CE/CME Course
Number analyzed (Participants) | 48
units on a scale | 8.9 (1.6)

5. Secondary Outcome: Perceived Course Relevance: Importance of Knowledge About Non-pharmacological Approaches
Description: Investigator-generated scale of perceived importance and relevance of course content: "How important is it for palliative care providers to know about non-pharmacological approaches to symptom management?" Likert scale ranges from 1 (not at all) to 4 (extremely).
Time Frame: 30 day follow-up
Population: There was missing data for one subject for this item.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Online CE/CME Course
Number analyzed (Participants) | 48
units on a scale | 3.9 (0.33)

6. Secondary Outcome: Perceived Course Relevance: Increasing Knowledge of Non-pharmacological Approaches
Description: Investigator-generated scale of perceived importance and relevance of course content: "How relevant is the content of this course for increasing palliative care providers' knowledge of non-pharmacological approaches?" Likert scale ranges from 1 (not at all) to 4 (extremely).
Time Frame: 30 day follow-up
Population: There was missing data for one subject for this item.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Online CE/CME Course
Number analyzed (Participants) | 48
units on a scale | 3.7 (0.59)

7. Secondary Outcome: Perceived Course Relevance: Potential of Course to Contribute to Improved Patient Care
Description: Investigator-generated scale of perceived importance and relevance of course content: "To what degree do you think this course could potentially contribute to improved patient care?" Likert scale ranges from 1 (not at all) to 4 (extremely).
Time Frame: 30 day follow-up
Population: There was missing data for one subject for this item.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Online CE/CME Course
Number analyzed (Participants) | 48
units on a scale | 3.5 (0.71)

ADVERSE EVENTS:
Description: Information on adverse events associated with this intervention was not solicited nor collected.
Groups:
- Online CE/CME Course: All subjects were assigned to take the three course modules of an online CE/CME course and complete pre- and post-course data collection. Module topics consisted of acupuncture, massage, and music-related interventions
Arm/Group | Online CE/CME Course
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No